CLINICAL TRIAL: NCT01216306
Title: Reducing Television Viewing To Prevent Obesity in Hispanic Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Jason Mendoza, Associate Professor of Pediatrics, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1K07CA131178 (NIH)
Record Dates: First submitted 2010-09-15; First posted 2010-10-07 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Obesity; Physical Activity; Sedentary Activity; Television Viewing
Keywords: Obesity; Physical Activity; Sedentary Activity; Television viewing; Latino; Hispanic; Preschool; School; Head Start
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Television reduction curriculum (Experimental): Students are taught the television reduction curriculum during the school day and parents are invited to attend after-school meetings to discuss reducing their children's television viewing.
  Interventions: Behavioral: Television reduction curriculum
- Control (No Intervention): Students will be taught the standard preschool curriculum.

INTERVENTIONS:
Behavioral: Television reduction curriculum — Students are taught the television reduction curriculum during the school day (15-30 minutes/day) 3-5 days/week over 7 weeks. Parents are invited to attend brief after-school meetings every other week to discuss reducing their children's television viewing.
  Other Names: Fit 5 Kids
  Arms: Television reduction curriculum

SUMMARY:
Obesity has been linked to the development of multiple cancers, and to poorer prognoses and higher mortality rates for certain pediatric and adult cancers. Preventing obesity is therefore a major strategy to prevent new cases of cancer and to decrease cancer related morbidity and mortality. In the US, childhood obesity is on the rise. Since childhood obesity strongly tracks into adulthood this epidemic among children greatly increases the risk of obesity and presumably cancer in adulthood. As a result, preventing childhood obesity has been selected as a major public health goal to reduce the risk and sequelae of obesity and cancer in the US.

Moreover, television (TV) viewing has been identified as a major risk factor for childhood obesity and US children spent more time watching TV than any other activity except sleep. TV viewing contributes to excess weight gain by decreasing physical activity and increasing caloric intake. The American Academy of Pediatrics (AAP) has issued national guidelines for parents to limit their children's total entertainment media time to no more than 1 to 2 hours of quality programming per day for children greater than 2 years of age. Low-income and minority children were at greater risk for exceeding this recommendation.

Few published interventions have been successful in decreasing TV viewing in children and only one was successful among preschool children. This intervention, "Fit 5 Kids" (i.e. fit by age 5 years), was a preschool curriculum designed to decrease TV viewing via age-appropriate lessons taught to the children by research staff. The curriculum also included a take-home component consisting of a newsletter with ideas for parent (for this grant, defined as the adult most responsible for the child's care, usually the mother) and child activities that complemented the school lesson plans. Although most behavioral interventions for preschoolers target parents rather than children, this curriculum was one of the few successful interventions targeted directly at children. However, Fit 5 Kids was not designed for or evaluated among Hispanic preschool children, the subpopulation of preschool children most severely affected by obesity. Moreover, no published intervention has successfully reduced both TV viewing and excess weight gain in any preschool population. In order to fill this gap, the investigators propose to evaluate a culturally adapted Fit 5 Kids TV reduction curriculum among Hispanic preschool children enrolled in the Head Start Program.

Fit 5 Kids is the TV reduction component of the Brocodile the Crocodile health promotion program. The overall goal of Fit 5 Kids is to teach the preschoolers to decrease their TV watching and encourage alternative activities such as family meals and active playtime. The primary goal of this research plan will be to conduct a pilot group randomized controlled trial evaluating the effectiveness of the adapted curriculum to reduce TV viewing and excess weight gain in low income, Hispanic preschool children

To achieve the project goals, the investigators Specific Aim includes:

1. To successfully recruit forty-eight 3-5 year old Hispanic children from 4 Head Start centers each year for 3 years and conduct a group randomized controlled study of the adapted Fit 5 Kids curriculum to evaluate its effectiveness in reducing TV viewing and excess weight gain in Hispanic preschool children.

The Primary Hypothesis to be tested includes:

H1. The culturally adapted Fit 5 Kids curriculum will reduce TV viewing and excess weight gain among Hispanic preschool children.

ELIGIBILITY:
Inclusion Criteria:

* 3-5 year old Hispanic children enrolled at the specific Head Start centers who have agreed to collaborate on this study

Exclusion Criteria:

* Clinically underweight, undernutrition, or failure to thrive

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 252 (Actual)
Dates: Start 2010-10; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Television viewing at follow up | The follow up measurement of television viewing will occur 8-10 weeks after the start of the study
  Television viewing (hours) will be measured by television viewing diaries completed by the parents for up to 7-days

SECONDARY OUTCOMES:
Adiposity and obesity at follow up | The follow up measurement of television viewing will occur 8-10 weeks after the start of the study
  Body mass index calculated from measured height and weight obtained per standard protocol. Waist circumference measured per standard protocol.
Physical activity at follow up | The follow up measurement of television viewing will occur 8-10 weeks after the start of the study
  Physical activity (duration and intensity) objectively measured by accelerometers for up to 7-days.

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Mendoza, MD, MPH, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Derived] Ogren M, Baranowski T, Lowry SJ, Mendoza JA. Model of goal directed behavior for limiting Latino preschoolers' television viewing: validity and reliability. BMC Public Health. 2020 Feb 5;20(1):185. doi: 10.1186/s12889-020-8268-x. PMID 32024491
- [Derived] Mendoza JA, Baranowski T, Jaramillo S, Fesinmeyer MD, Haaland W, Thompson D, Nicklas TA. Fit 5 Kids TV Reduction Program for Latino Preschoolers: A Cluster Randomized Controlled Trial. Am J Prev Med. 2016 May;50(5):584-592. doi: 10.1016/j.amepre.2015.09.017. Epub 2015 Nov 10. PMID 26572093